CLINICAL TRIAL: NCT04828980
Title: Impact of Different Virtual Reality Experiences on Anxiety and Pain
Brief Title: Utilization of Different Virtual Reality Experiences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Ryan Li, MD, Assistant Professor of Otolaryngology - Head and Neck Surgery, Division of Head and Neck Surgery, School of Medicine, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 00022194
Record Dates: First submitted 2021-03-28; First posted 2021-04-02 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Surgery; Pain, Postoperative; Anxiety; Otolaryngological Disease
MeSH Terms: conditions — Pain, Postoperative; Anxiety Disorders; Otorhinolaryngologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Virtual Reality Experience (Active Comparator): Patients will be provided with a mindfulness VR experience for use up to 15 minutes at bedside.
  Interventions: Device: Oculus Quest: TRIPP
- Gaming Virtual Reality Experience (Active Comparator): Patients will be provided with an active gaming VR experience for use up to 15 minutes at bedside.
  Interventions: Device: Oculus Quest: Angry Birds

INTERVENTIONS:
Device: Oculus Quest: TRIPP — This is a VR experience that focuses on meditation and mindfulness
  Arms: Mindfulness Virtual Reality Experience
Device: Oculus Quest: Angry Birds — This is an active gaming VR experience that utilizes controllers to aim and launch objects at targets.
  Arms: Gaming Virtual Reality Experience

SUMMARY:
This trial studies differences between a mindfulness and a gaming virtual reality (VR) experience as a means for preoperative anxiety management and postoperative pain management among patients after head and neck surgery. Investigators will assess differences in anxiety scores, pain scores, physiologic measures, and subjective patient experiences.

DETAILED DESCRIPTION:
Optimal postoperative pain control after head and neck surgery is vital for recovery, and non-pharmacologic strategies to improve pain may help reduce narcotic use. Further, preoperative anxiety is common and can impact postoperative pain, analgesic requirements, and recovery. In addition to facilitating with postoperative pain control, VR may have a role in reducing preoperative anxiety. However, it is unclear whether different VR experiences may be more beneficial for different clinical applications.

This study will evaluate if there are differences in preoperative anxiety and postoperative pain when utilizing different VR experiences. Patients undergoing head and neck surgery will be randomly allocated preoperatively to first participate in either a mindfulness or active gaming VR experience, and then postoperatively will crossover and participate in the other experience they did not utilize prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing head and neck surgery
* Are able to provide informed consent

Exclusion Criteria:

* Isolation precautions
* Active eye discharge
* Active nausea or vomiting
* History of seizure, epilepsy, or hypersensitivity to flashing light
* Expected to have wounds or wound care that prevent comfortable and safe use of the VR headset

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
Change in patient-reported anxiety | baseline, and then 15 minutes later after VR use
  Anxiety level will be obtained using a 100mm Visual Analogue Scale (VAS). Preoperative anxiety scores will be obtained prior to VR then immmediately after VR use to assess change in anxiety after each intervention. Score will range from 0 (no anxiety) to 100 (extremely anxious)
Change in patient-reported pain | baseline, and then 15 minutes later after VR use
  Pain level will be obtained using a 100mm Visual Analogue Scale (VAS). Postoperative pain scores will be obtained prior to VR then immmediately after VR use to assess change in pain level after each intervention. Score will range from 0 (no pain) to 100 (worst pain imaginable)

SECONDARY OUTCOMES:
Change in blood pressure | baseline, and then 15 minutes later after VR use
  Blood pressure (mmHG) will be recorded prior to VR use and then after VR use to assess change in physiologic responses after each intervention.
Patient experience | 1 minute after use of VR
  Patients will complete a short survey at the completion of their participation in each VR experience evaluating their experience using a 5-point Likert scale, with responses ranging from 1 (low satisfaction) to 5 (high satisfaction)
Change in heart rate | baseline, and then 15 minutes later after VR use
  Heart rate (beats per minute [bpm]) will be recorded prior to VR use and then after VR use to assess change in physiologic responses after each intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Li, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No